CLINICAL TRIAL: NCT02302742
Title: PROspective Evaluation of GErmline Mutations, Cancer Outcome and Tissue Biomarkers: A Registry for Patients With Triple Negative Breast Cancer and Germline Mutations
Brief Title: Triple Negative Breast Cancer and Germline Hereditary Breast and Ovarian Cancer Mutation Carrier Registry
Acronym: PROGECT
Status: Recruiting | Type: Observational
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, Priyanka Sharma, Professor of Medicine, University of Kansas
Other Study IDs: KUMC 12614
Record Dates: First submitted 2014-11-11; First posted 2014-11-27 (Estimated); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer; Hereditary Breast and Ovarian Cancer
Keywords: Triple Negative Breast Cancer; TNBC; Hereditary Breast and Ovarian Cancer; HBOC; Prospective Registry
MeSH Terms: conditions — Breast Neoplasms; Hereditary Breast and Ovarian Cancer Syndrome; Triple Negative Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — A baseline blood draw is collected as a part of this registry. If a study participant has a personal history of cancer and a tumor sample is available, the participant may give consent for the tissue to be used as a part of the study. Additional optional specimen collection sub-studies may also be offered to participants.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Triple Negative Breast Cancer patients: No intervention
- Germline HBOC Mutation Carriers: No intervention

SUMMARY:
PROGECT is a registry for patients with Triple Negative breast cancer (TNBC) or patients who have an identified germline mutations (such as a mutation on the BRCA1 or BRCA2 genes).

DETAILED DESCRIPTION:
This study is being done to collect cancer-related information from patients with triple negative breast cancer and patients with hereditary genetic mutations. This information will help us better understand the link between genetic changes and cancer outcome in patients with triple negative breast cancer.

ELIGIBILITY:
Inclusion criteria include:

Triple Negative Breast Cancer

* ER/PR <10% and HER negative per current ASCO/CAP guidelines
* Stages I-IV
* Any age at diagnosis
* Patient must be within 5 years of diagnosis
* Eligible regardless of genetic testing status
* Genetic testing recommended for patients meeting NCCN and Medicare guidelines

AND/OR

Germline mutation Carriers

* Patients with deleterious or uncertain mutations in HBOC genes (BRCA, PTEN, P53, -PALB2 etc) are eligible regardless of type/site of cancer
* Healthy patients harboring mutations also eligible
* There is no time limit from the time of diagnosis of cancer and enrollment.
* Eligible regardless of personal history of cancer

Exclusion Criteria include:

Triple Negative Breast Cancer -Patient is not within five years of diagnosis

Germline mutation Carriers:

-Patient only carries a HBOC mutation that is classified as "polymorphism" of "favor polymorphism"

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Academic Center & Community Clinics
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2011-03-22 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Prevalence of germline mutations (such as BRCA1/2 mutations) in patients with TNBC | 5 years
. Predictors of response to neo/adjuvant chemotherapy in patients with TNBC | 5 years
Long term Disease free and overall survival rates in TNBC patients treated with different systemic therapies | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Priyanka Sharma, MD, Principal Investigator — University of Kansas Medical Center
Locations (11):
- United States (11):
  - Hays Medical Center Dreiling-Schmidt Cancer Institute, Hays, Kansas
  - KCCC West, Kansas City, Kansas
  - KCCC Overland Park, Overland Park, Kansas
  - Overland Park Regional Medical Center, Overland Park, Kansas
  - Salina Regional Health Center - Tammy Walker Cancer Center, Salina, Kansas
  - The University of Kansas Cancer Center, Westwood, Kansas
  - Universtiy Health, Kansas City, Missouri
  - KCCC South, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - KCCC - North, Kansas City, Missouri
  - KCCC Lee's Summit, Lee's Summit, Missouri

REFERENCES:
- [Background] Sharma P, Klemp JR, Kimler BF, Mahnken JD, Geier LJ, Khan QJ, Elia M, Connor CS, McGinness MK, Mammen JM, Wagner JL, Ward C, Ranallo L, Knight CJ, Stecklein SR, Jensen RA, Fabian CJ, Godwin AK. Germline BRCA mutation evaluation in a prospective triple-negative breast cancer registry: implications for hereditary breast and/or ovarian cancer syndrome testing. Breast Cancer Res Treat. 2014 Jun;145(3):707-14. doi: 10.1007/s10549-014-2980-0. Epub 2014 May 7. PMID 24807107
- [Background] Connor CS, Kimler BF, Mammen JM, McGinness MK, Wagner JL, Alsop SM, Ward C, Fabian CJ, Khan QJ, Sharma P. Impact of neoadjuvant chemotherapy on axillary nodal involvement in patients with clinically node negative triple negative breast cancer. J Surg Oncol. 2015 Feb;111(2):198-202. doi: 10.1002/jso.23790. Epub 2014 Sep 29. PMID 25266871